CLINICAL TRIAL: NCT04339491
Title: What Are the Factors That Affect the Physical Activity Levels of Young Adults During Social Isolation Due to Coronavirus?
Brief Title: Physical Activity During Social Isolation
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Saliha Gürdal Karakelle, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 30042020-1
Record Dates: First submitted 2020-04-03; First posted 2020-04-09 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Social Isolation
Keywords: physical activity; young adult; coronavirus
MeSH Terms: conditions — Social Isolation; Motor Activity; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to evaluate the physical activity level and the factors affecting physical activity among young adults who are socially isolated due to coronavirus.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-50
* Being volunteer

Exclusion Criteria:

* Being unable to communicate in Turkish
* Not knowing read and write in Turkish

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young Adults from Community Sample
Sampling Method: Probability Sample
Enrollment: 1206 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Exercise Habit and Factors Affecting Exercise Attendance | The assessment will be made once at baseline, data collection will be completed up to 6 weeks.
  It was created by the researchers due to the fact that the existing surveys could not meet the pandemic period. It will be questioned whether the participants had exercise habits in the times before the pandemic. Possible reasons will be questioned according to the positive and negative answers. The answers of the questions are yes / no and they will not be scored. Frequency evaluation will be made according to the results obtained.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire - Short Form (IPAQ-SF) | The assessment will be made once at baseline, data collection will be completed up to 6 weeks.
  IPAQ-SF provides information on walking, moderate and vigorous activities and time spent sitting, within a week. There are two forms of output from scoring the IPAQ. Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity.
Exercise Benefits/Barriers Scale | The assessment will be made once at baseline, data collection will be completed up to 6 weeks.
  It was developed in response to a need for an instrument to determine perceptions of individuals concerning the benefits and barriers to participating in exercise. The scale, which is a 4-point Likert type, has 4 responses from 4 (strongly agree) to 1 (strongly disagree). The total score of the scale varies between 43-172. Higher scores mean that knowing the benefits of exercise and no barrier to exercise.
The Pittsburgh Sleep Quality Index | The assessment will be made once at baseline, data collection will be completed up to 6 weeks.
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. It consists of 24 questions, 18 of which are included in the scoring. Each question is scored between 0-3 and the highest total score is 21. The high total score indicates poor sleep quality.
The Hospital Anxiety and Depression Scale | The assessment will be made once at baseline, data collection will be completed up to 6 weeks.
  A self-assessment scale has been developed and found to be a reliable instrument for detecting states of depression and anxiety. The questions of the scale, which is a 4-point Likert type, are scored between 0-3. The total score is obtained between 0-21. The high score indicates the presence of depression and anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Zengin Alpözgen, PhD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Özge Ertan, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No